CLINICAL TRIAL: NCT06954051
Title: Validation of Game-based Assessment of Emotion Regulation Abilities Using the REThink Life Online Game in a Population of Adolescents and Young Adults
Brief Title: ERFs Game-based Assessment in AYAs: Validation of Game-based Assessment of Emotion Regulation Abilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Oana David, Professor PhD, Babes-Bolyai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REThinkRESILIENT
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Emotion Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REThink Life (Other): The participants will complete the scale measurements after receiving the four levels of the REThink Life game, each focusing on an emotion regulation skill and an associated assessment system.
  Interventions: Other: REThink Life

INTERVENTIONS:
Other: REThink Life — REThink Life is a therapeutic game developed by David and collaborators (2019) and it is composed of four levels, each training a different emotion regulation ability (emotion recognition, mindfulness, distinguishing between rational and irrational thoughts, and positive attention bias).

SUMMARY:
This activity will have the objective of establishing the validity of in-game emotion regulation abilities assessment for adolescents and young adults.

DETAILED DESCRIPTION:
Each level of the REThink LIFE online game dedicated to training a specific ER skill has an assessment task for emotion recognition, stress reactivity, mindfulness and positive attention abilities. The aim of this study will be to investigate the validity of in-game performance measurements or scores as indicators of adolescents and young adults' emotion regulation abilities.

ELIGIBILITY:
Inclusion Criteria:

* adolescents and young adults with between 10 and 24 years old provided with written parental consent where applicable

Exclusion Criteria:

* intellectual disability or physical limitations precluded the use of the computer program

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 230 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Emotion regulation | Baseline
  The Cognitive Emotion Regulation Questionnaire (CERQ-short) is an 18-item scale assessing nine different emotion regulation strategies, namely Self-blame, Other-blame, Rumination, Catastrophizing, Positive refocusing, Planning, Positive reappraisal, Putting into perspective and Acceptance. Children and adolescents were asked to express the frequency of using each strategy on a 5-point Likert-type scale, from 1 ("almost never") to 5 ("almost always"). Higher scores on adaptive strategies (e.g., positive reappraisal, refocus on planning, positive refocusing, putting into perspective, acceptance) are equivalent to a better outcome (more adaptive coping). Higher scores on maladaptive strategies (e.g., rumination, catastrophizing, self-blame, other-blame) are equivalent to worse outcomes (less adaptive coping).
Behavioral difficulties | Baseline
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioural screening questionnaire for children aged 2 to 17 years old, encompassing emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior.
  Total difficulties score: Sum of all subscales except Prosocial → Range: 0 to 40. Prosocial score is reported separately → Range: 0 to 10. Higher scores on total difficulties and the four problem subscales are equivalent to worse outcomes. Higher scores on the prosocial subscale are equivalent to better outcomes.
Stress | Baseline
  The Adolescent Stress Scale (ADOSS) will be used to capture students' level of stress in the following domains: personal, academic, family, and social. Total score ranges from 20 to 100, with higher scores indicating higher levels of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Oana A. David, Ph.D, Principal Investigator — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No